CLINICAL TRIAL: NCT03475394
Title: Comparison of Effectiveness of Morus Alba and Chlorhexidine Gels on Moderate Periodontitis Among 35 to 55 Year Old Subjects: A Hospital Based Randomized Controlled Trial
Brief Title: Effectiveness of Locally Delivered Morus Alba Gel on Moderate Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLE VK Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr. Shilpa Gunjal, Associate Professor, KLE VK Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLEU/Ethic/14-15/D-79
Record Dates: First submitted 2018-03-15; First posted 2018-03-23 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Chronic Periodontitis
Keywords: Chlorhexidine gluconate; Morus alba; Microbiology; Gel; Root planing
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Chlorhexidine gel) (Active Comparator): Non surgical periodontal treatment at baseline and 0.1 ml of 1% chlorhexidine gel administered in subsequent visits.
  Interventions: Other: Chlorhexidine gel
- Group 2 (Morus alba gel) (Experimental): Non surgical periodontal treatment at baseline and 0.1 ml of 16% Morus alba gel administered in subsequent visits.
  Interventions: Other: Morus alba gel
- Group 3 (Placebo) (Placebo Comparator): Non surgical periodontal treatment at baseline and 0.1 ml of placebo gel administered in subsequent visits.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Chlorhexidine gel — 0.1 ml of Chlorhexidine gel was administered into the periodontal pocket
  Arms: Group 1 (Chlorhexidine gel)
Other: Morus alba gel — 0.1 ml of Morus alba gel was administered into the periodontal pocket
  Arms: Group 2 (Morus alba gel)
Other: Placebo — 0.1 ml of Placebo gel was administered into the periodontal pocket
  Arms: Group 3 (Placebo)

SUMMARY:
Background: Periodontitis is a chronic inflammatory disease of tooth and supporting tissues with clinical signs of bone and connective tissue loss and is mediated by a combination of periodontal pathogens and host defense systems. Currently the use of herbal products in dentistry is increasing due to their easy availability, low cost and lesser side effects. One such herbal plant is Morus alba which is known to possess medicinal properties. Therefore the present study was conducted to determine the clinical effectiveness of subgingivally delivered Morus alba gel incorporated into polaxamers vehicle for its controlled release on periodontal pocket in adjunct to scaling and root planing for treatment of moderate periodontitis patients.

Methods: one hundred eighty patients with chronic periodontitis having pocket depth of ≥5 mm in atleast two different teeth were treated by full-mouth scaling and root planning (SRP) and curettage. They were randomly assigned into one of the three groups with 60 in each group: Group 1: Chlorhexidine Sol-gel was applied at baseline, 15 and 30 days. Group 2: Morus alba Sol-gel was applied at baseline, 15 and 30 days. Grpup 3: Placebo gel was applied at baseline, 15 and 30 days. Plaque index (PI) (Silness and Loe), Gingival index (GI) (Loe and Silness), Community Periodontal index, Periodontal pocket depth and quantitative analysis (anaerobic culture) of Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis and Tannerella forsythia were assessed at baseline and after 45 days.

DETAILED DESCRIPTION:
Morus alba is invaluable member of the plant kingdom belonging to the family Moraceae and the genus Morus. It is extensively cultivated for leaf yield in sericulture. Morus alba have long been used in traditional medicine to improve eyesight, lower blood pressure, prevent diabetes, protect the liver, strengthen joints and treat fever. In particular, few studies on mulberry fruits have reported its biological activities such as antioxidative and anti-inflammatory activities. Even the root bark of has been traditionally used in Asian countries for medicinal purposes due to its anti-inflammatory, hypoglycemic, antibacterial activities. LD50 of extracts of Morus Alba leaves was found to be above 2000 mg/kg which is safe to be used in human beings. Therefore, in the present study the Morus alba leaves has been used in the gel preparation and its effectiveness is assessed against periodontal microorganisms.

ELIGIBILITY:
Inclusion Criteria:

1. 35 to 55 years old
2. untreated moderate chronic periodontitis having probing pocket depth of ≥5 mm in atleast two different teeth

Exclusion Criteria:

1. use of antibiotics or anti-inflammatory drugs during the last 6 months before baseline examination
2. Received periodontal treatment in the last 6 months
3. pregnant or lactating
4. allergy to chlorhexidine or any of the components in the tested products
5. using tobacco products in any form
6. systemic diseases (e.g., diabetes mellitus, hypertension and immunological disorders)
7. ) orthodontic treatment
8. alcoholics
9. removable prostheses
10. Healthy with a normal BMI

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the periodontal pocket depth | 45 days
  Measured by Probing pocket depth

SECONDARY OUTCOMES:
Reduction in the Microbial count of periodontal pathogens | 45 days
  Reduction in Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis and Tannerella forsythia
Reduction in Plaque deposition | 45 days
  Measured by Plquel index (Silness and Loe)
Reduction in gingival inflammation | 45 days
  Measured by Gingival index (Loe and Silness)

IPD SHARING:
Plan to Share IPD: No